CLINICAL TRIAL: NCT00981968
Title: An Investigator- And Subjects- Blind Phase 1 Study To Investigate Pharmacokinetics, Safety And Tolerability Of Sitaxentan In Japanese Healthy Subjects Following Single And Multiple Doses And Western Healthy Subjects Following Single Dose
Brief Title: Phase 1, Single and Multiple Doses Study of Sitaxentan in Japanese and Western Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B1321046
Record Dates: First submitted 2009-09-21; First posted 2009-09-22 (Estimated); Last update posted 2010-10-15 (Estimated); Status verified 2010-10

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Japanese Cohort (Experimental): Single and multiple oral doses of sitaxentan sodium or placebo in 12 healthy subjects.
  Interventions: Drug: Sitaxentan sodium/Placebo
- Western Cohort (Experimental): Single oral dose of sitaxentan sodium in 10 healthy subjects.
  Interventions: Drug: Sitaxentan sodium/Placebo

INTERVENTIONS:
Drug: Sitaxentan sodium/Placebo — 100 mg and 200 mg, tablet, single and multiple oral doses for 7 days
  Other Names: Thelin
  Arms: Japanese Cohort
Drug: Sitaxentan sodium/Placebo — 100 mg and 200 mg, tablet, single oral dose
  Other Names: Thelin
  Arms: Western Cohort

SUMMARY:
The purpose of this study is to investigate safety, tolerability and pharmacokinetics of sitaxentan following single and multiple oral administrations of sitaxentan sodium in Japanese healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

Healthy male and/or female subjects between the age of 18 and 55 years, inclusive.

Body Mass Index of 17.5 to 33.5 kg/m2, and a total body weight >45 kg. Mean body weight and the body weight range of Western subjects are similar to those of Japanese subjects with a 10% plus and minus error.

Exclusion Criteria:

Pregnant or nursing females; females of childbearing potential who are unwilling or unable to use an acceptable method of contraception.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2009-09; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Adverse events (spontaneous and solicited) | Day 0 to Day 9 of Period 3 for cohort 1, Day 0 to Day 3 of Period 2 for cohort 2
ECGs, Vital signs, Safety laboratory test | Screening visit to Day 9 of Period 3 for cohort 1 and Day 3 of Period 2 for cohort 2
Pharmacokinetics (single dose): Cmax, Tmax, AUC, t1/2, CL/F and V/F | Day 1 of Periods 1 and 2
Pharmacokinetics (multiple dose): Cmax, Tmax, Ctrough, AUC, t1/2, CL/F, V/F, Rac and Rss | Days 1 and 7 of Periods 1 and 3

SECONDARY OUTCOMES:
No secondary outcome | No secondary outcome

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Glendale, California, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1321046&StudyName=Phase%201%2C%20single%20and%20multiple%20doses%20study%20of%20sitaxentan%20in%20Japanese%20and%20Western%20subjects